CLINICAL TRIAL: NCT02487394
Title: Protein Biomarker Discovery and Validation in COPD And Asthma
Brief Title: Protein Biomarker Discovery and Validation in Chronic Obstructive Pulmonary Disease (COPD) And Asthma
Acronym: Proteomics
Status: Terminated | Type: Observational
Why Stopped: NIH Funded Grant Expired
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 13-0462
Record Dates: First submitted 2015-02-12; First posted 2015-07-01 (Estimated); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- COPD Smoker Subjects: Smokers Active smoking will be defined as daily use of cigarettes, pipes, cigarillos or cigars at time of entry into the study and through duration of study.
  Interventions: Procedure: Exhaled Breath Condensate (EBC)
- Asthma Non-Smoker Subjects: Non-Smokers Subjects with no active smoking. No active smoking defined as never smoking or having stopped smoking for 5 years or greater.
  Interventions: Procedure: Exhaled Breath Condensate (EBC)

INTERVENTIONS:
Procedure: Exhaled Breath Condensate (EBC) — Collection of EBC condensate

SUMMARY:
The purpose of the study is to better understand proteomics of asthma and COPD, and response to therapy. There are two Phases to this study broken into two arms. In Phase I, we propose is to use discovery proteomics and techniques to identify protein expression signatures. Subjects who complete Phase I are eligible, but not required, to enroll in Phase II. In Phase II, we propose to establish and validate the predictive value of protein signatures for treatment responses using inhaled corticosteroids.

DETAILED DESCRIPTION:
There are two Phases to this study broken into two arms. In Phase I, our propose to use discovery proteomics and high throughput techniques to identify protein expression signatures. The total planned size of Phase I is 100 patients. Patients will be divided into two arms based on disease status (COPD or asthma). Active smoking will be defined as daily use of cigarettes, pipes, cigarillos or cigars at time of entry into the study and through duration of study. No active smoking defined as never smoking or having stopped smoking for 5 years or greater.

In the Phase II, we aim to establish and validate the predictive value of proteomic signatures for therapeutic responses using inhaled corticosteroids. For Phase II, subjects who completed Phase I are eligible, but not required to participate in Phase II.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for Asthma

INCLUSION

* History consistent with asthma: episodic wheezing, shortness of breath, or cough
* Airway lability recognized by at least 12% improvement in Forced Expiratory Volume (FEV1) after 2 puffs of beta2 agonist Age >18yrs
* FEV1 >40% predicted
* Never smoker, current smoker, or quit smoking ≥5 years ago Criteria for COPD

INCLUSION

* History consistent with COPD: dyspnea with exertion, productive cough, progressive course
* Smoking history of at least 20 pack years
* Current smoker or quit smoking ≥5 years ago
* Age >18yrs
* FEV1: Forced Vital Capacity (FVC) ratio < 0.70 following 2 puffs of albuterol
* FEV1 greater than 50% predicted

Exclusion Criteria:

* Exclusion for Asthma EXCLUSION

  * Other respiratory illness other than asthma
  * Chronic infectious process
  * Significant other medical illness
  * Inability to consent
  * Pregnancy Exclusion for COPD EXCLUSION
  * Other respiratory illness other than COPD
  * Chronic infectious process
  * Significant other medical illness
  * Inability to consent
  * Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be divided into two identical arms based on smoking status. One arm will contain subjects who are active smokers and the other arm will contain subjects with no active smoking.
  Each arm will contain 50 subjects, 26 with COPD (Stage II and III with 13 subjects in each) along with 24 asthmatics (Mild to Moderate disease with 12 subjects in each).
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Calhoun, M.D., Principal Investigator — UTMB
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Anticipated to enroll both smoking and non-smoking asthma subjects. Anticipated to enroll both smoking and non-smoking COPD subjects. NO smoking asthmatic subjects enrolled. NO non-smoking COPD subjects enrolled. There are only two groups.
Groups:
- Asthma Subjects-Non-Smokers: Asthma subjects were required to have a phyician diagnosis of asthma, requiring as needed beta2 agonists, with or without an inhaled corticosteroid.
  No smoking asthmatic subjects were included in this arm.
- COPD Subjects-Smokers: COPD subjects were required to have a physician diagnosis of COPD, and treatment with short- or long-acting muscarinic antagonists, or short- or long-acting beta2 agonists, with or without inhaled corticosteroids. All COPD subjects were current smokers. We did not enroll former smokers in this arm.
Period: Phase 1
Arm/Group | Asthma Subjects-Non-Smokers | COPD Subjects-Smokers
Started | 8 | 1
Completed (One subject was withdrawn) | 8 | 0
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Phase 2
Arm/Group | Asthma Subjects-Non-Smokers | COPD Subjects-Smokers
Started (Only 4 subjects who completed phase I enrolled in phase II of asthmatics. None of the COPD subjects who completed phase 1 enrolled in phase II.) | 4 | 0
Completed | 4 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The overall participants was a total of 9.
Groups:
- Asthma, Non-Smokers: No active smoking defined as never smoking or having stopped smoking for 5 years or greater.
- COPD, Smokers: Active smoking will be defined as daily use of cigarettes, pipes, cigarillos or cigars at time of entry into the study and through duration of study.
- Total: Total of all reporting groups
Arm/Group | Asthma, Non-Smokers | COPD, Smokers | Total
Number analyzed (Participants) | 8 | 1 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 1 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 6
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 8 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Exhaled Breath Condensate Protein Concentration
Description: Protein concentrations were below the limit of detectability and are not scientifically robust.
Time Frame: 1 year through study completion
Population: An observational Study principally for collecting biological samples.
Measure: Median (Standard Deviation); unit: ug/ml
Groups:
- COPD, Smokers: For Phase II, Phase II will again be divided into two arms based on active smoking status as discussed previously.
  Asthma, Smokers and Non-Smokers: Comparing protein expressions between the two groups.
  COPD, Smokers and Non-Smokers: We will validate the prdictive value of the proteomic signatures for therapeutic responses.
- Asthma, Non-Smokers: In Phase I, One arm will contain subjects who are active smokers and the other arm will contain subjects with no active smoking. Active smoking will be defined as daily use of cigarettes, pipes, cigarillos or cigars at time of entry into the study and through duration of study. No active smoking defined as never smoking or having stopped smoking for 5 years or greater.
  Asthma, Smokers and Non-Smokers: Comparing protein expressions between the two groups.
  COPD, Smokers and Non-Smokers: We will validate the prdictive value of the proteomic signatures for therapeutic responses.
Arm/Group | COPD, Smokers | Asthma, Non-Smokers
Number analyzed (Participants) | 1 | 8
ug/ml | NA (0) — All concentrations below the level of detection | NA (0) — All concentrations below the level of detection

ADVERSE EVENTS:
Groups:
- Asthma, Non-Smokers: Asthma subjects were required to have a phyician diagnosis of asthma, requiring PRN beta2 agonists, with or without an inhaled corticosteroid.
  No smoking asthmatic subjects were included in this arm.
- COPD, Smokers: COPD subjects were required to have a physician diagnosis of COPD, and treatment with short- or long-acting muscarinic antagonists, or short- or long-acting beta2 agonists, with or without inhaled corticosteroids. All COPD subjects were current smokers. We did not enroll former smokers in this arm.
Arm/Group | Asthma, Non-Smokers | COPD, Smokers
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/1
Other Adverse Events (participants affected / at risk) | 0/8 | 0/1

LIMITATIONS AND CAVEATS:
It was anticipated to enroll in 4 arms of the study, only 2 arms had successful enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No